CLINICAL TRIAL: NCT01061736
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter, Two-part, Dose Ranging and Confirmatory Study With an Operationally Seamless Design, Evaluating Efficacy and Safety of SAR153191 on Top of Methotrexate (MTX) in Patients With Active Rheumatoid Arthritis Who Are Inadequate Responders to MTX Therapy
Brief Title: Evaluation of Sarilumab (SAR153191/REGN88) on Top of Methotrexate in Rheumatoid Arthritis Patients
Acronym: RA-MOBILITY
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EFC11072; 2009-016266-90 (EudraCT Number)
Record Dates: First submitted 2010-02-02; First posted 2010-02-03 (Estimated); Results first posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — sarilumab; Methotrexate; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (10):
- Part A: SAR 100 mg qw (Experimental): Sarilumab 100 mg subcutaneous (SC) injection weekly (qw) on top of MTX for 12 weeks.
  Interventions: Drug: Sarilumab; Drug: Methotrexate; Drug: Folic Acid
- Part A: SAR 150 mg qw (Experimental): Sarilumab 150 mg SC injection qw on top of MTX for 12 weeks.
  Interventions: Drug: Sarilumab; Drug: Methotrexate; Drug: Folic Acid
- Part A: SAR 100 mg q2w (Experimental): Sarilumab 100 mg SC injection every other week (q2w) alternating with placebo on top of MTX for 12 weeks.
  Interventions: Drug: Sarilumab; Drug: Placebo (for sarilumab); Drug: Methotrexate; Drug: Folic Acid
- Part A: SAR 150 mg q2w (Experimental): Sarilumab 150 mg SC injection q2w alternating with placebo on top of MTX for 12 weeks.
  Interventions: Drug: Sarilumab; Drug: Placebo (for sarilumab); Drug: Methotrexate; Drug: Folic Acid
- Part A: SAR 200 mg q2w (Experimental): Sarilumab 200 mg SC injection q2w alternating with placebo on top of MTX for 12 weeks.
  Interventions: Drug: Sarilumab; Drug: Placebo (for sarilumab); Drug: Methotrexate; Drug: Folic Acid
- Part A: Placebo qw (Placebo Comparator): Placebo (for sarilumab) qw on top of MTX for 12 weeks.
  Interventions: Drug: Placebo (for sarilumab); Drug: Methotrexate; Drug: Folic Acid
- Part B Cohort 1: Non-selected Doses (Experimental): Sarilumab 100 mg qw, 150 mg qw or 100 mg q2w SC injections as in Part A on top of MTX up to dose selection. After dose selection, participants were not continued but were allowed to participate in the open-label, long-term, extension study SARIL-RA-EXTEND (LTS11210).
  Interventions: Drug: Sarilumab; Drug: Placebo (for sarilumab); Drug: Methotrexate; Drug: Folic Acid
- Part B: SAR 150 mg q2w (Cohort 1[Selected Dose]+Cohort 2) (Experimental): Sarilumab 150 mg SC injection q2w on top of MTX for a maximum of 52 weeks. Participants with inadequate response from Week 16 could be rescued with open-label highest dose of sarilumab.
  Interventions: Drug: Sarilumab; Drug: Methotrexate; Drug: Folic Acid
- Part B: SAR 200 mg q2w (Cohort 1[Selected Dose]+Cohort 2) (Experimental): Sarilumab 200 mg SC injection q2w on top of MTX for a maximum of 52 weeks. Participants with inadequate response from Week 16 could be rescued with open-label highest dose of sarilumab.
  Interventions: Drug: Sarilumab; Drug: Methotrexate; Drug: Folic Acid
- Part B: Placebo q2w (Cohort 1[Selected Dose]+Cohort 2) (Experimental): Placebo (for sarilumab) q2w on top of MTX for a maximum of 52 weeks. Participants with inadequate response from Week 16 could be rescued with open-label highest dose of sarilumab.
  Interventions: Drug: Placebo (for sarilumab); Drug: Methotrexate; Drug: Folic Acid

INTERVENTIONS:
Drug: Sarilumab — Pharmaceutical form: solution for injection
  Route of administration: subcutaneous
  Other Names: SAR153191; REGN88
  Arms: Part A: SAR 100 mg q2w; Part A: SAR 100 mg qw; Part A: SAR 150 mg q2w; Part A: SAR 150 mg qw; Part A: SAR 200 mg q2w; Part B Cohort 1: Non-selected Doses; Part B: SAR 150 mg q2w (Cohort 1[Selected Dose]+Cohort 2); Part B: SAR 200 mg q2w (Cohort 1[Selected Dose]+Cohort 2)
Drug: Placebo (for sarilumab) — Pharmaceutical form: solution for injection
  Route of administration: subcutaneous
  Arms: Part A: Placebo qw; Part A: SAR 100 mg q2w; Part A: SAR 150 mg q2w; Part A: SAR 200 mg q2w; Part B Cohort 1: Non-selected Doses; Part B: Placebo q2w (Cohort 1[Selected Dose]+Cohort 2)
Drug: Methotrexate — Same weekly dose as received prior to enrollment
Drug: Folic Acid — According to local standard

SUMMARY:
Primary Objectives:

Part A (dose ranging study):

To demonstrate that sarilumab (SAR153191/REGN88) on top of MTX was effective on reduction of signs and symptoms of rheumatoid arthritis at 12 weeks.

Part B (pivotal study):

To demonstrate that sarilumab added to MTX was effective in:

* reduction of signs and symptoms of rheumatoid arthritis at 24 weeks
* inhibition of progression of structural damage at 52 weeks
* improvement in physical function at 16 weeks

Secondary Objectives:

Part B:

To demonstrate that sarilumab added to MTX was effective in induction of a major clinical response at 52 weeks

To assess the safety of sarilumab added to MTX

To document the pharmacokinetic profile of sarilumab added to MTX in participants with active rheumatoid arthritis who were inadequate responders to MTX therapy.

DETAILED DESCRIPTION:
The total study duration for a participant was 16-22 weeks (Part A) and 56-62 weeks (Part B) broken down as follows:

* Screening: Up to 4 weeks
* Treatment: 12 weeks (Part A) and 52 weeks (Part B)*
* Follow-up: 6 weeks (for participants who would not continue in the long-term extension study).

'*' Participants successfully completing their treatment period would be offered the opportunity to enter the long term extension study LTS11210 (SARIL-RA-EXTEND) (NCT01146652).

ELIGIBILITY:
Inclusion criteria :

* Diagnosis of rheumatoid arthritis ≥3 months duration
* Active disease defined as:

  * at least 8/68 tender joints and 6/66 swollen joints,
  * high sensitivity C-reactive protein (hs-CRP) >6 mg/l,
  * continuous treatment with MTX for at least 12 weeks prior to baseline visit and on stable dose for at least 6 weeks prior to screening visit.

Part B only:

* Bone erosion based on documented X-ray prior to first study drug intake, or
* Cyclic Citrullinated Peptide (CCP) positive, or
* Rheumatoid Factor (RF) positive.

Exclusion criteria:

* Age <18 years or >75 years.
* Treatment with disease-modifying antirheumatic drugs (DMARDs) other than MTX within 4 weeks or 12 weeks prior to screening (depending on DMARDs).
* Past history of non-response to prior Tumor Necrosis Factor (TNF) or biologic treatment.
* Any past or current biologic agents for the treatment of rheumatoid arthritis within 3 months.
* Use of parenteral glucocorticoids or intraarticular glucocorticoids within 4 weeks prior to screening visit.
* Use of oral glucocorticoid greater than 10mg/day or equivalent/day, or a change in dosage within 4 weeks prior to baseline visit.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1675 (Actual)
Dates: Start 2010-03; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark C Genovese, MD, Professor of Medicine, Principal Investigator — Division of Immunology and Rheumatology - Stanford University - USA; TWJ Huizinga, Prof Dr, Study Chair — Dpt of Rheumatology - Leiden University Medical Center - The Netherlands
Locations (262):
- United States (45):
  - Investigational Site Number 840070, Anniston, Alabama
  - Investigational Site Number 840004, Birmingham, Alabama
  - Investigational Site Number 840072, Gilbert, Arizona
  - Investigational Site Number 840029, Beverly Hills, California
  - Investigational Site Number 840007, Palm Desert, California
  - Investigational Site Number 840008, San Francisco, California
  - Investigational Site Number 840021, Santa Maria, California
  - Investigational Site Number 840049, Upland, California
  - Investigational Site Number 840050, Dunedin, Florida
  - Investigational Site Number 840041, Jacksonville, Florida
  - Investigational Site Number 840067, Jupiter, Florida
  - Investigational Site Number 840048, Miami, Florida
  - Investigational Site Number 840006, Orlando, Florida
  - Investigational Site Number 840063, Palm Harbor, Florida
  - Investigational Site Number 840060, Sarasota, Florida
  - Investigational Site Number 840003, Atlanta, Georgia
  - Investigational Site Number 840028, Decatur, Georgia
  - Investigational Site Number 840027, Marietta, Georgia
  - Investigational Site Number 840018, Idaho Falls, Idaho
  - Investigational Site Number 840046, Chicago, Illinois
  - Investigational Site Number 840015, Lexington, Kentucky
  - Investigational Site Number 840073, Cumberland, Maryland
  - Investigational Site Number 840055, Frederick, Maryland
  - Investigational Site Number 840013, Wheaton, Maryland
  - Investigational Site Number 840066, St Louis, Missouri
  - Investigational Site Number 840071, Omaha, Nebraska
  - Investigational Site Number 840056, New York, New York
  - Investigational Site Number 840068, Hickory, North Carolina
  - Investigational Site Number 840044, Toledo, Ohio
  - Investigational Site Number 840002, Oklahoma City, Oklahoma
  - Investigational Site Number 840011, Tulsa, Oklahoma
  - Investigational Site Number 840065, Tulsa, Oklahoma
  - Investigational Site Number 840010, Bethlehem, Pennsylvania
  - Investigational Site Number 840009, Duncansville, Pennsylvania
  - Investigational Site Number 840062, Reading, Pennsylvania
  - Investigational Site Number 840058, Columbia, South Carolina
  - Investigational Site Number 840016, North Charleston, South Carolina
  - Investigational Site Number 840025, Jackson, Tennessee
  - Investigational Site Number 840001, Dallas, Texas
  - Investigational Site Number 840022, Dallas, Texas
  - Investigational Site Number 840012, Dallas, Texas
  - Investigational Site Number 840020, Houston, Texas
  - Investigational Site Number 840069, Lubbock, Texas
  - Investigational Site Number 840074, Mesquite, Texas
  - Investigational Site Number 840061, Tacoma, Washington
- Argentina (12):
  - Investigational Site Number 032005, Buenos Aires
  - Investigational Site Number 032007, Buenos Aires
  - Investigational Site Number 032008, Buenos Aires
  - Investigational Site Number 032006, Caba
  - Investigational Site Number 032002, Córdoba
  - Investigational Site Number 032003, Córdoba
  - Investigational Site Number 032012, Mar del Plata
  - Investigational Site Number 032011, Quilmes
  - Investigational Site Number 032010, Ramos Mejía
  - Investigational Site Number 032001, Rosario
  - Investigational Site Number 032004, San Miguel de Tucumán
  - Investigational Site Number 032009, Zárate
- Australia (12):
  - Investigational Site Number 036003, Camperdown
  - Investigational Site Number 036005, Clayton
  - Investigational Site Number 036012, Fitzroy
  - Investigational Site Number 036010, Garran
  - Investigational Site Number 036004, Heidelberg West
  - Investigational Site Number 036009, Herston
  - Investigational Site Number 036002, Malvern East
  - Investigational Site Number 036001, Maroochydore
  - Investigational Site Number 036006, St Leonards
  - Investigational Site Number 036011, Sydney
  - Investigational Site Number 036014, Victoria Park
  - Investigational Site Number 036007, Woodville
- Austria (2):
  - Investigational Site Number 040001, Graz
  - Investigational Site Number 040002, Vienna
- Belarus (2):
  - Investigational Site Number 112002, Minsk
  - Investigational Site Number 112001, Minsk
- Belgium (2):
  - Investigational Site Number 056003, Genk
  - Investigational Site Number 056001, Liège
- Brazil (11):
  - Investigational Site Number 076008, Campinas
  - Investigational Site Number 076012, Campinas
  - Investigational Site Number 076001, Curitiba
  - Investigational Site Number 076006, Goiânia
  - Investigational Site Number 076010, Juiz de Fora
  - Investigational Site Number 076004, Porto Alegre
  - Investigational Site Number 076005, Rio de Janeiro
  - Investigational Site Number 076011, Salvador
  - Investigational Site Number 076002, São Paulo
  - Investigational Site Number 076003, São Paulo
  - Investigational Site Number 076013, Vitória
- Canada (7):
  - Investigational Site Number 124004, Burlington
  - Investigational Site Number 124003, Mississauga
  - Investigational Site Number 124008, Newmarket
  - Investigational Site Number 124002, St. Catharines
  - Investigational Site Number 124005, Toronto
  - Investigational Site Number 124001, Toronto
  - Investigational Site Number 124012, Winnipeg
- Chile (13):
  - Investigational Site Number 152005, Osorno
  - Investigational Site Number 152010, Port Montt
  - Investigational Site Number 152012, Santiago
  - Investigational Site Number 152001, Santiago
  - Investigational Site Number 152002, Santiago
  - Investigational Site Number 152008, Santiago
  - Investigational Site Number 152009, Santiago
  - Investigational Site Number 152011, Santiago
  - Investigational Site Number 152013, Santiago
  - Investigational Site Number 152014, Talca
  - Investigational Site Number 152004, Valdivia
  - Investigational Site Number 152007, Viña del Mar
  - Investigational Site Number 152006, Viña del Mar
- Colombia (8):
  - Investigational Site Number 170004, Barranquilla
  - Investigational Site Number 170001, Bogotá
  - Investigational Site Number 170003, Bogotá
  - Investigational Site Number 170006, Bogotá
  - Investigational Site Number 170008, Bogotá
  - Investigational Site Number 170007, Bucaramanga
  - Investigational Site Number 170009, Bucaramanga
  - Investigational Site Number 170002, Medellín
- Czechia (4):
  - Investigational Site Number 203005, Brno
  - Investigational Site Number 203004, Hlučín
  - Investigational Site Number 203001, Prague
  - Investigational Site Number 203002, Uherské Hradiště
- Egypt (2):
  - Investigational Site Number 818001, Cairo
  - Investigational Site Number 818002, Cairo
- Estonia (2):
  - Investigational Site Number 233001, Tallinn
  - Investigational Site Number 233002, Tallinn
- Finland (3):
  - Investigational Site Number 246001, Helsinki
  - Investigational Site Number 246002, Hyvinkää
  - Investigational Site Number 246003, Pori
- Germany (10):
  - Investigational Site Number 276007, Berlin
  - Investigational Site Number 276008, Berlin
  - Investigational Site Number 276004, Erlangen
  - Investigational Site Number 276003, Frankfurt am Main
  - Investigational Site Number 276015, Halle
  - Investigational Site Number 276005, Hamburg
  - Investigational Site Number 276013, Hamburg
  - Investigational Site Number 276012, Heidelberg
  - Investigational Site Number 276001, Herne
  - Investigational Site Number 276006, Hildesheim
- Greece (3):
  - Investigational Site Number 300001, Athens
  - Investigational Site Number 300002, Heraklion
  - Investigational Site Number 300003, Thessaloniki
- Hungary (9):
  - Investigational Site Number 348006, Budapest
  - Investigational Site Number 348014, Budapest
  - Investigational Site Number 348003, Debrecen
  - Investigational Site Number 348010, Debrecen
  - Investigational Site Number 348011, Eger
  - Investigational Site Number 348013, Gy?r
  - Investigational Site Number 348005, Sátoraljaújhely
  - Investigational Site Number 348015, Szombathely
  - Investigational Site Number 348004, Veszprém
- India (12):
  - Investigational Site Number 356015, Ahmedabad
  - Investigational Site Number 356007, Bangalore
  - Investigational Site Number 356003, Chennai
  - Investigational Site Number 356012, Hyderabad
  - Investigational Site Number 356005, Hyderabad
  - Investigational Site Number 356011, Lucknow
  - Investigational Site Number 356013, Lucknow
  - Investigational Site Number 356001, Maharashtra
  - Investigational Site Number 356010, Mumbai
  - Investigational Site Number 356004, Mumbai
  - Investigational Site Number 356002, New Delhi
  - Investigational Site Number 356008, New Delhi
- Lithuania (2):
  - Investigational Site Number 440001, Kaunas
  - Investigational Site Number 440002, Vilnius
- Malaysia (3):
  - Investigational Site Number 458001, Ipoh
  - Investigational Site Number 458002, Kuching
  - Investigational Site Number 458003, Putrajaya
- Mexico (8):
  - Investigational Site Number 484008, Durango
  - Investigational Site Number 484002, Guadalajara
  - Investigational Site Number 484007, Metepec
  - Investigational Site Number 484001, Mexico City
  - Investigational Site Number 484003, Mexico City
  - Investigational Site Number 484004, Mérida
  - Investigational Site Number 484009, Mérida
  - Investigational Site Number 484005, Monterrey
- Investigational Site Number 528002, Heerlen, Netherlands
- New Zealand (4):
  - Investigational Site Number 554004, Christchurch
  - Investigational Site Number 554002, Rotorua
  - Investigational Site Number 554003, Tauranga
  - Investigational Site Number 554001, Timaru
- Norway (2):
  - Investigational Site Number 578004, Kristiansand
  - Investigational Site Number 578006, Tønsberg
- Philippines (3):
  - Investigational Site Number 608003, Cebu City
  - Investigational Site Number 608001, Manila
  - Investigational Site Number 608002, Manila
- Poland (7):
  - Investigational Site Number 616002, Bialystok
  - Investigational Site Number 616003, Bialystok
  - Investigational Site Number 616001, Krakow
  - Investigational Site Number 616005, Lublin
  - Investigational Site Number 616006, Torun
  - Investigational Site Number 616004, Warsaw
  - Investigational Site Number 616012, Wroclaw
- Portugal (3):
  - Investigational Site Number 620003, Aveiro
  - Investigational Site Number 620001, Lisbon
  - Investigational Site Number 620002, Lisbon
- Romania (8):
  - Investigational Site Number 642006, Brăila
  - Investigational Site Number 642001, Bucharest
  - Investigational Site Number 642002, Bucharest
  - Investigational Site Number 642003, Bucharest
  - Investigational Site Number 642004, Bucharest
  - Investigational Site Number 642010, Bucharest
  - Investigational Site Number 642005, Galati
  - Investigational Site Number 642008, Ploieşti
- Russia (15):
  - Investigational Site Number 643017, Kemerovo
  - Investigational Site Number 643006, Kemerovo
  - Investigational Site Number 643004, Moscow
  - Investigational Site Number 643020, Moscow
  - Investigational Site Number 643001, Moscow
  - Investigational Site Number 643002, Moscow
  - Investigational Site Number 643012, Moscow
  - Investigational Site Number 643009, Novosibirsk
  - Investigational Site Number 643016, Ryazan
  - Investigational Site Number 643007, Saint Petersburg
  - Investigational Site Number 643008, Saint Petersburg
  - Investigational Site Number 643014, Saint Petersburg
  - Investigational Site Number 643010, Samara
  - Investigational Site Number 643011, Saratov
  - Investigational Site Number 643013, Ufa
- South Africa (11):
  - Investigational Site Number 710011, Cape Town
  - Investigational Site Number 710007, Cape Town
  - Investigational Site Number 710009, Cape Town
  - Investigational Site Number 710003, Durban
  - Investigational Site Number 710002, Durban
  - Investigational Site Number 710001, Johannesburg
  - Investigational Site Number 710004, Kempton Park
  - Investigational Site Number 710005, Pretoria
  - Investigational Site Number 710006, Pretoria
  - Investigational Site Number 710008, Pretoria
  - Investigational Site Number 710010, Stellenbosch
- South Korea (14):
  - Investigational Site Number 410014, Anyang
  - Investigational Site Number 410006, Busan
  - Investigational Site Number 410004, Daegu
  - Investigational Site Number 410013, Daegu
  - Investigational Site Number 410005, Daejeon
  - Investigational Site Number 410010, Gwangju
  - Investigational Site Number 410009, Incheon
  - Investigational Site Number 410001, Incheon
  - Investigational Site Number 410011, Jeonju
  - Investigational Site Number 410007, Seoul
  - Investigational Site Number 410012, Seoul
  - Investigational Site Number 410003, Seoul
  - Investigational Site Number 410002, Seoul
  - Investigational Site Number 410008, Suwon
- Spain (5):
  - Investigational Site Number 724009, A Coruña
  - Investigational Site Number 724010, Barcelona
  - Investigational Site Number 724011, Sabadell
  - Investigational Site Number 724012, Santiago de Compostela
  - Investigational Site Number 724007, Seville
- Taiwan (2):
  - Investigational Site Number 158002, Linkou District
  - Investigational Site Number 158001, Taipei
- Thailand (2):
  - Investigational Site Number 764001, Bangkok
  - Investigational Site Number 764003, Bangkok
- Turkey (Türkiye) (5):
  - Investigational Site Number 792003, Adana
  - Investigational Site Number 792002, Ankara
  - Investigational Site Number 792005, Ankara
  - Investigational Site Number 792004, Antalya
  - Investigational Site Number 792001, Izmir
- Ukraine (8):
  - Investigational Site Number 804003, Dnipropetrovsk
  - Investigational Site Number 804002, Donetsk
  - Investigational Site Number 804010, Kharkiv
  - Investigational Site Number 804008, Kyiv
  - Investigational Site Number 804004, Kyiv
  - Investigational Site Number 804005, Lviv
  - Investigational Site Number 804006, Simferopol
  - Investigational Site Number 804009, Zaporizhzhia

REFERENCES:
- [Background] Strand V, Kosinski M, Chen CI, Joseph G, Rendas-Baum R, Graham NM, van Hoogstraten H, Bayliss M, Fan C, Huizinga T, Genovese MC. Sarilumab plus methotrexate improves patient-reported outcomes in patients with active rheumatoid arthritis and inadequate responses to methotrexate: results of a phase III trial. Arthritis Res Ther. 2016 Sep 6;18(1):198. doi: 10.1186/s13075-016-1096-9. PMID 27600829
- [Result] Huizinga TW, Fleischmann RM, Jasson M, Radin AR, van Adelsberg J, Fiore S, Huang X, Yancopoulos GD, Stahl N, Genovese MC. Sarilumab, a fully human monoclonal antibody against IL-6Ralpha in patients with rheumatoid arthritis and an inadequate response to methotrexate: efficacy and safety results from the randomised SARIL-RA-MOBILITY Part A trial. Ann Rheum Dis. 2014 Sep;73(9):1626-34. doi: 10.1136/annrheumdis-2013-204405. Epub 2013 Dec 2. PMID 24297381
- [Result] Genovese MC, Fleischmann R, Kivitz AJ, Rell-Bakalarska M, Martincova R, Fiore S, Rohane P, van Hoogstraten H, Garg A, Fan C, van Adelsberg J, Weinstein SP, Graham NM, Stahl N, Yancopoulos GD, Huizinga TW, van der Heijde D. Sarilumab Plus Methotrexate in Patients With Active Rheumatoid Arthritis and Inadequate Response to Methotrexate: Results of a Phase III Study. Arthritis Rheumatol. 2015 Jun;67(6):1424-37. doi: 10.1002/art.39093. PMID 25733246
- [Derived] Choy E, Bykerk V, Lee YC, van Hoogstraten H, Ford K, Praestgaard A, Perrot S, Pope J, Sebba A. Disproportionate articular pain is a frequent phenomenon in rheumatoid arthritis and responds to treatment with sarilumab. Rheumatology (Oxford). 2023 Jul 5;62(7):2386-2393. doi: 10.1093/rheumatology/keac659. PMID 36413080
- [Derived] Rubbert-Roth A, Furst DE, Fiore S, Praestgaard A, Bykerk V, Bingham CO, Charles-Schoeman C, Burmester G. Association between low hemoglobin, clinical measures, and patient-reported outcomes in patients with rheumatoid arthritis: results from post hoc analyses of three phase III trials of sarilumab. Arthritis Res Ther. 2022 Aug 25;24(1):207. doi: 10.1186/s13075-022-02891-x. PMID 36008838
- [Derived] Rehberg M, Giegerich C, Praestgaard A, van Hoogstraten H, Iglesias-Rodriguez M, Curtis JR, Gottenberg JE, Schwarting A, Castaneda S, Rubbert-Roth A, Choy EHS; MOBILITY, MONARCH, TARGET, and ASCERTAIN investigators. Identification of a Rule to Predict Response to Sarilumab in Patients with Rheumatoid Arthritis Using Machine Learning and Clinical Trial Data. Rheumatol Ther. 2021 Dec;8(4):1661-1675. doi: 10.1007/s40744-021-00361-5. Epub 2021 Sep 14. PMID 34519964
- [Derived] Genovese MC, Burmester GR, Hagino O, Thangavelu K, Iglesias-Rodriguez M, John GS, Gonzalez-Gay MA, Mandrup-Poulsen T, Fleischmann R. Interleukin-6 receptor blockade or TNFalpha inhibition for reducing glycaemia in patients with RA and diabetes: post hoc analyses of three randomised, controlled trials. Arthritis Res Ther. 2020 Sep 9;22(1):206. doi: 10.1186/s13075-020-02229-5. PMID 32907617
- [Derived] Genovese MC, Fleischmann R, Kivitz A, Lee EB, van Hoogstraten H, Kimura T, St John G, Mangan EK, Burmester GR. Efficacy and safety of sarilumab in combination with csDMARDs or as monotherapy in subpopulations of patients with moderately to severely active rheumatoid arthritis in three phase III randomized, controlled studies. Arthritis Res Ther. 2020 Jun 10;22(1):139. doi: 10.1186/s13075-020-02194-z. PMID 32522251
- [Derived] Boyapati A, Schwartzman S, Msihid J, Choy E, Genovese MC, Burmester GR, Lam G, Kimura T, Sadeh J, Weinreich DM, Yancopoulos GD, Graham NMH. Association of High Serum Interleukin-6 Levels With Severe Progression of Rheumatoid Arthritis and Increased Treatment Response Differentiating Sarilumab From Adalimumab or Methotrexate in a Post Hoc Analysis. Arthritis Rheumatol. 2020 Sep;72(9):1456-1466. doi: 10.1002/art.41299. Epub 2020 Aug 25. PMID 32343882
- [Derived] Genovese MC, van der Heijde D, Lin Y, St John G, Wang S, van Hoogstraten H, Gomez-Reino JJ, Kivitz A, Maldonado-Cocco JA, Seriolo B, Stanislav M, Burmester GR. Long-term safety and efficacy of sarilumab plus methotrexate on disease activity, physical function and radiographic progression: 5 years of sarilumab plus methotrexate treatment. RMD Open. 2019 Aug 1;5(2):e000887. doi: 10.1136/rmdopen-2018-000887. eCollection 2019. PMID 31452928
- [Derived] Muszbek N, Proudfoot C, Fournier M, Chen CI, Kuznik A, Kiss Z, Gal P, Michaud K. Economic Evaluation of Sarilumab in the Treatment of Adult Patients with Moderately-to-Severely Active Rheumatoid Arthritis Who Have an Inadequate Response to Conventional Synthetic Disease-Modifying Antirheumatic Drugs. Adv Ther. 2019 Jun;36(6):1337-1357. doi: 10.1007/s12325-019-00946-1. Epub 2019 Apr 19. PMID 31004324
- [Derived] Boyapati A, Msihid J, Fiore S, van Adelsberg J, Graham NM, Hamilton JD. Sarilumab plus methotrexate suppresses circulating biomarkers of bone resorption and synovial damage in patients with rheumatoid arthritis and inadequate response to methotrexate: a biomarker study of MOBILITY. Arthritis Res Ther. 2016 Oct 6;18(1):225. doi: 10.1186/s13075-016-1132-9. PMID 27716324

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 247 centers in 36 countries. Overall, 3715 participants were screened between March 2010 and July 2012, 2040 of whom were screen failures. Screen failures were mainly due to failure to meet the inclusion criterion for severity of the disease and/or due to meeting the exclusion criterion.
Pre-assignment Details: Randomization was performed centrally with allocation generated by Interactive Voice/Web Response System, stratified by geographical region and prior biological use. 306 participants were randomized in Part A. 1369 participants were randomized in part B, 172 before dose selection (cohort 1) and 1197 after dose selection (cohort 2).
Groups:
- Part A: SAR 100 mg qw: Sarilumab 100 mg subcutaneous (SC) injection weekly (qw) on top of methotrexate (MTX) for 12 weeks.
- Part B: SAR 150 mg q2w (Cohort 1 [Selected Dose]+Cohort 2): Sarilumab 150 mg SC injection q2w on top of MTX for a maximum of 52 weeks. Participants with inadequate response from Week 16 could be rescued with high dose of sarilumab (SAR 200 mg q2w).
- Part B: SAR 200 mg q2w (Cohort 1 [Selected Dose]+Cohort 2): Sarilumab 200 mg SC injection q2w on top of MTX for a maximum of 52 weeks. Participants with inadequate response from Week 16 could be rescued with high dose of sarilumab (SAR 200 mg q2w).
- Part B: Placebo q2w (Cohort 1[Selected Dose]+Cohort 2): Placebo (for sarilumab) q2w on top of MTX for a maximum of 52 weeks. Participants with inadequate response from Week 16 could be rescued with high dose of sarilumab (SAR 200 mg q2w).
Period: Overall Study
Arm/Group | Part A: SAR 100 mg qw | Part A: SAR 150 mg qw | Part A: SAR 100 mg q2w | Part A: SAR 150 mg q2w | Part A: SAR 200 mg q2w | Part A: Placebo qw | Part B Cohort 1: Non-selected Doses | Part B: SAR 150 mg q2w (Cohort 1 [Selected Dose]+Cohort 2) | Part B: SAR 200 mg q2w (Cohort 1 [Selected Dose]+Cohort 2) | Part B: Placebo q2w (Cohort 1[Selected Dose]+Cohort 2)
Started | 50 | 50 | 51 | 51 | 52 | 52 | 84 | 430 | 427 | 428
Treated | 50 | 50 | 51 | 51 | 51 | 52 | 84 | 428 | 426 | 428
Rescued | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 61 (Included both participants who completed and did not complete the study.) | 55 (Included both participants who completed and did not complete the study.) | 168 (Included both participants who completed and did not complete the study.)
Completed | 37 | 46 | 45 | 48 | 45 | 49 | 0 | 336 | 330 | 354
Not Completed | 13 | 4 | 6 | 3 | 7 | 3 | 84 | 94 | 97 | 74
Not completed — Dose regimen not selected | 0 | 0 | 0 | 0 | 0 | 0 | 79 | 0 | 0 | 0
Not completed — Adverse Event | 13 | 1 | 3 | 2 | 4 | 1 | 4 | 63 | 67 | 34
Not completed — Lack of Efficacy | 0 | 2 | 1 | 1 | 1 | 2 | 1 | 9 | 9 | 10
Not completed — Poor compliance to protocol | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 5 | 9
Not completed — Not treated | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0
Not completed — Other than specified above | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 18 | 15 | 21

BASELINE CHARACTERISTICS:
Groups:
- Part A: SAR 100 mg qw: Sarilumab 100 mg SC injection qw on top of MTX for 12 weeks.
- Part A: SAR 100 mg q2w: Sarilumab 100 mg SC injection q2w alternating with placebo on top of MTX for 12 weeks.
- Part B Cohort 1: Non-selected Doses: Sarilumab 100 mg qw, 150 mg qw or 100 mg q2w SC injections on top of MTX up to dose selection. After dose selection, participants were not continued but were allowed to participate in the open-label, long-term, extension study SARIL-RA-EXTEND (LTS11210).
- Part B: SAR 150 mg q2w (Cohort 1[Selected Dose]+Cohort 2): Sarilumab 150 mg SC injection q2w on top of MTX for a maximum of 52 weeks. Participants with inadequate response from Week 16 could be rescued with high dose of sarilumab (SAR 200 mg q2w).
- Part B: SAR 200 mg q2w (Cohort 1[Selected Dose]+Cohort 2): Sarilumab 200 mg SC injection q2w on top of MTX for a maximum of 52 weeks. Participants with inadequate response from Week 16 could be rescued with high dose of sarilumab (SAR 200 mg q2w).
- Total: Total of all reporting groups
Arm/Group | Part A: SAR 100 mg qw | Part A: SAR 150 mg qw | Part A: SAR 100 mg q2w | Part A: SAR 150 mg q2w | Part A: SAR 200 mg q2w | Part A: Placebo qw | Part B Cohort 1: Non-selected Doses | Part B: SAR 150 mg q2w (Cohort 1[Selected Dose]+Cohort 2) | Part B: SAR 200 mg q2w (Cohort 1[Selected Dose]+Cohort 2) | Part B: Placebo q2w (Cohort 1[Selected Dose]+Cohort 2) | Total
Number analyzed (Participants) | 50 | 50 | 51 | 51 | 52 | 52 | 84 | 430 | 427 | 428 | 1675
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (12.3) | 50.9 (11.1) | 53.5 (11.8) | 51.2 (12.9) | 48.7 (12.4) | 55.2 (12.5) | 51.1 (11.5) | 50.3 (11.9) | 50.8 (12.0) | 51.1 (11.2) | 51.04 (11.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 42 | 38 | 42 | 42 | 38 | 69 | 345 | 359 | 346 | 1362
  Male | 9 | 8 | 13 | 9 | 10 | 14 | 15 | 85 | 68 | 82 | 313

OUTCOME MEASURES:

1. Primary Outcome: Part A: Percentage of Participants Achieving American College of Rheumatology 20% (ACR20) Response at Week 12
Description: ACR20 response was defined, based on guidelines set forth by the American College of Rheumatology (ACR), as ≥20 % improvement in tender joint count and swollen joint count as well as ≥20% improvement in at least 3 of 5 following measures: C-Reactive Protein (CRP), Participant assessment of pain; Participant's global assessment of disease activity; Physician global assessment of disease activity; and Health Assessment Question-Disability Index (HAQ-DI). Missing data imputed by Last Observation Carried Forward (LOCF).
Time Frame: Baseline to Week 12
Population: Part A Intent-to-treat (ITT) population defined as all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Part A: SAR 100 mg qw | Part A: SAR 150 mg qw | Part A: SAR 100 mg q2w | Part A: SAR 150 mg q2w | Part A: SAR 200 mg q2w | Part A: Placebo qw
Number analyzed (Participants) | 50 | 50 | 51 | 51 | 52 | 52
Percentage of participants | 62 | 72 | 49 | 66.7 | 65.4 | 46.2
Statistical Analysis 1: Comparison: Part A: SAR 100 mg qw vs Part A: Placebo qw; Analysis was performed using two-sided Cochran-Mantel-Haenszel test. Pairwise comparisons of the response rates between each dose of sarilumab and placebo were derived. The multiplicity issues were addressed by using the Hommel-procedure; Test type: Superiority or Other; p = 0.1155, Cochran-Mantel-Haenszel — Threshold for significance = 0.05; Odds Ratio (OR) = 1.99, 95% CI 2-sided [0.85 to 4.64]
Statistical Analysis 2: Comparison: Part A: SAR 150 mg qw vs Part A: Placebo qw; Test type: Superiority or Other; p = 0.0041, Cochran-Mantel-Haenszel — Threshold for significance = 0.05; Odds Ratio (OR) = 3.84, 95% CI 2-sided [1.53 to 9.63]
Statistical Analysis 3: Comparison: Part A: SAR 100 mg q2w vs Part A: Placebo qw; Test type: Superiority or Other; p = 0.7119, Cochran-Mantel-Haenszel — Threshold for significance = 0.05; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.52 to 2.61]
Statistical Analysis 4: Comparison: Part A: SAR 150 mg q2w vs Part A: Placebo qw; Test type: Superiority or Other; p = 0.0363, Cochran-Mantel-Haenszel — Threshold for significance = 0.05; Odds Ratio (OR) = 2.38, 95% CI 2-sided [1.06 to 5.35]
Statistical Analysis 5: Comparison: Part A: SAR 200 mg q2w vs Part A: Placebo qw; Test type: Superiority or Other; p = 0.0426, Cochran-Mantel-Haenszel — Threshold for significance = 0.05; Odds Ratio (OR) = 2.34, 95% CI 2-sided [1.03 to 5.29]

2. Primary Outcome: Part B: Percentage of Participants Achieving ACR20 Response at Week 24
Description: ACR20 improvement responses were determined without imputation of missing post-baseline values. In addition data collected after treatment discontinuation or rescue was set to missing. Responder status was determined if possible. With these rules, participants automatically became non-responders for all time points beyond the time point they started rescue treatment or discontinued study treatment.
Time Frame: Baseline to Week 24
Population: ITT population which included all participants randomized after dose selection (cohort 2).
Measure: Number; unit: Percentage of participants
Groups:
- Part B: SAR 150 mg q2w: Participants randomized after dose selection received Sarilumab 150 mg SC injection q2w on top of MTX for a maximum of 52 weeks.
- Part B: SAR 200 mg q2w: Participants randomized after dose selection received Sarilumab 200 mg SC injection q2w on top of MTX for a maximum of 52 weeks.
- Part B: Placebo q2w: Participants randomized after dose selection received Placebo (for sarilumab) q2w on top of MTX for a maximum of 52 weeks
Arm/Group | Part B: SAR 150 mg q2w | Part B: SAR 200 mg q2w | Part B: Placebo q2w
Number analyzed (Participants) | 400 | 399 | 398
Percentage of participants | 58 | 66.4 | 33.4
Statistical Analysis 1: Comparison: Part B: SAR 150 mg q2w vs Part B: Placebo q2w; Analysis was performed using two-sided Cochran-Mantel-Haenszel test. Pairwise comparisons of the response rates between each dose of sarilumab and placebo was derived. The multiplicity issues for part B were addressed by using a Bonferroni correction for each dose together with a hierarchical testing procedure across the 3 co-primary and the main secondary endpoints. The hierarchical testing sequence continued only when previous endpoint was statistically significant at 0.025 level; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance = 0.025; Odds Ratio (OR) = 2.773, 95% CI 2-sided [2.077 to 3.703]
Statistical Analysis 2: Comparison: Part B: SAR 200 mg q2w vs Part B: Placebo q2w; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance = 0.025; Odds Ratio (OR) = 3.975, 95% CI 2-sided [2.957 to 5.344]

3. Primary Outcome: Part B: Change From Baseline in Health Assessment Question Disability Index (HAQ-DI) at Week 16
Description: HAQ-DI was a participant-reported questionnaire that assesses the difficulty of performing daily activities: dress/groom, arise, eat, walk, reach, grip, hygiene and common activities. Overall score range from 0=least difficulty to 3=extreme difficulty. An increase in the score indicates a worsening of physical function while a decrease in the score represents improvement. Data collected after treatment discontinuation was set to missing.
Time Frame: Baseline, Week 16
Population: Cohort 2 ITT population only and included participants with available data of HAQ-DI at baseline and on or before Week 16.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part B: SAR 150 mg q2w | Part B: SAR 200 mg q2w | Part B: Placebo q2w
Number analyzed (Participants) | 362 | 365 | 378
units on a scale
  Baseline | 1.63 (0.63) | 1.69 (0.63) | 1.61 (0.65)
  Week 16 | 1.08 (0.67) | 1.11 (0.7) | 1.31 (0.67)
  Change from baseline at Week 16 | -0.54 (0.55) | -0.58 (0.63) | -0.3 (0.58)
Statistical Analysis 1: Comparison: Part B: SAR 150 mg q2w vs Part B: Placebo q2w; Analysis was performed using a mixed model for repeated measures (MMRM). Differences in least square (LS) mean between each dose of sarilumab and placebo were derived. Testing was performed according to the hierarchical testing procedure (performed only when the previous endpoint was statistically significant); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance = 0.025; LS mean difference = -0.235, 95% CI 2-sided [-0.312 to -0.157]
Statistical Analysis 2: Comparison: Part B: SAR 200 mg q2w vs Part B: Placebo q2w; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance = 0.025; LS mean difference = -0.258, 95% CI 2-sided [-0.336 to -0.181]

4. Primary Outcome: Part B: Change From Baseline in Van Der Heijde Modified Total Sharp Score (mTSS) at Week 52
Description: The Sharp method modified by D. van der Heijde involves separate scores for erosions and joint space narrowing based on radiographs to assess the degree of structural damage. Total score range from 0 (normal) to 448 (worst possible total score). An increase in total score represents progression of structural damage. Missing data were imputed by the linear extrapolation method.
Time Frame: Baseline, Week 52
Population: Cohort 2 ITT population and included participants with available data of mTSS at baseline and on or before Week 52.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part B: SAR 150 mg q2w | Part B: SAR 200 mg q2w | Part B: Placebo q2w
Number analyzed (Participants) | 352 | 359 | 352
units on a scale
  Baseline | 54.67 (63.42) | 46.34 (57.43) | 48.01 (65.23)
  Week 52 | 55.57 (63.73) | 46.59 (57.63) | 50.79 (65.82)
  Change from baseline at Week 52 | 0.90 (4.66) | 0.25 (4.61) | 2.78 (7.73)
Statistical Analysis 1: Comparison: Part B: SAR 150 mg q2w vs Part B: Placebo q2w; Analysis was performed using two-sided rank-based ANCOVA model. Testing was performed according to the hierarchical testing procedure (performed only when the previous endpoints were statistically significant); Test type: Superiority or Other; p < 0.0001, Rank ANCOVA — Threshold for significance = 0.025
Statistical Analysis 2: Comparison: Part B: SAR 200 mg q2w vs Part B: Placebo q2w; Test type: Superiority or Other; p < 0.0001, Rank ANCOVA — Threshold for significance = 0.025

5. Secondary Outcome: Part B: Percentage of Participants Achieving a Major Clinical Response at Week 52
Description: Major clinical response was defined as an ACR70 response maintained for at least 24 consecutive weeks. ACR70 response uses the same criteria as for ACR20 but requires 70% improvement. In the primary approach, data collected after treatment discontinuation or rescue was set to missing. No imputation of missing post-baseline values was performed. Responder status was determined if possible. With these rules, participants automatically became non-responders for all time points beyond the time point they started rescue treatment or discontinued study treatment.
Time Frame: Baseline up to Week 52
Population: ITT population which included all participants randomized after dose selection (cohort 2).
Measure: Number; unit: Percentage of participants
Arm/Group | Part B: SAR 150 mg q2w | Part B: SAR 200 mg q2w | Part B: Placebo q2w
Number analyzed (Participants) | 400 | 399 | 398
Percentage of participants | 12.8 | 14.8 | 3
Statistical Analysis 1: Comparison: Part B: SAR 150 mg q2w vs Part B: Placebo q2w; Analysis was performed using two-sided Cochran-Mantel-Haenszel test. Pairwise comparisons of the response rates between each dose of sarilumab and placebo were derived. Testing was performed according to the hierarchical testing procedure (performed only when the previous endpoints were statistically significant); Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance = 0.025; Odds Ratio (OR) = 4.661, 95% CI 2-sided [2.451 to 8.863]
Statistical Analysis 2: Comparison: Part B: SAR 200 mg q2w vs Part B: Placebo q2w; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance = 0.025; Odds Ratio (OR) = 5.565, 95% CI 2-sided [2.946 to 10.515]

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to study completion regardless of seriousness or relationship to investigational medicinal product (IMP).
Description: Reported adverse events are treatment-emergent adverse events that is AEs that developed/worsened during the 'on treatment period' (from the first IMP injection up to the end of the study). Safety population defined as all randomized participants who received at least one dose of IMP.
Groups:
- Part A: SAR 100 mg qw: Part A participants exposed to sarilumab 100 mg qw on top of MTX (mean exposure of 10 weeks).
- Part A: SAR 150 mg qw: Part A participants exposed to sarilumab 150 mg qw on top of MTX (mean exposure of 12 weeks).
- Part A: SAR 100 mg q2w: Part A participants exposed to sarilumab 100 mg q2w on top of MTX (mean exposure of 11 weeks).
- Part A: SAR 150 mg q2w: Part A participants exposed to sarilumab 150 mg q2w on top of MTX (mean exposure of 12 weeks). Included the participant randomized to placebo qw who received sarilumab 150 mg q2w in error.
- Part A: SAR 200 mg q2w: Part A participants exposed to sarilumab 200 mg q2w on top of MTX (mean exposure of 11 weeks).
- Part A: Placebo qw: Part A participants exposed to placebo on top of MTX (mean exposure of 12 weeks). Excluded 1 participant who received an erroneous IMP kit with sarilumab 150 mg q2w. He/she was considered in the 150 mg q2w treatment group for safety analysis.
- Part B: SAR 100 mg qw Cohort 1 (Non-selected Dose): Part B participants exposed to sarilumab 100 mg qw on top of MTX (mean exposure of 10 weeks).
- Part B: SAR 150 mg qw Cohort 1 (Non-selected Dose): Part B participants exposed to sarilumab 150 mg qw on top of MTX (mean exposure of 12 weeks). Excluded 1 participant who received sarilumab 100 mg q2w in error. He/she was considered in the 100 mg q2w treatment group for safety analysis.
- Part B: SAR 100 mg q2w Cohort 1 (Non-selected Dose): Part B participants exposed to sarilumab 100 mg q2w on top of MTX (mean exposure of 13 weeks). Included 1 participant who received sarilumab 100 mg q2w in error.
- Part B: SAR 150 mg q2w (Cohort 1[Selected Dose]+Cohort 2): Part B participants exposed to sarilumab 150 mg q2w on top of MTX (mean exposure of 42 weeks). 61 participants with inadequate response from Week 16 rescued with high dose of sarilumab (SAR 200 mg q2w) were not included. Included 3 participants randomized to sarilumab 200 mg q2w who received at least one dose of sarilumab 150 mg q2w in error.
- Part B: SAR 200 mg q2w (Cohort 1[Selected Dose]+Cohort 2): Part B participants exposed to sarilumab 200 mg q2w on top of MTX (mean exposure of 42 weeks). 55 participants with inadequate response from Week 16 rescued with high dose of sarilumab (SAR 200 mg q2w) were not included. Excluded 3 participants randomized to sarilumab 200 mg q2w who received at least one dose of sarilumab 150 mg q2w in error and included a participant randomized to placebo q2w who received sarilumab 200 mg q2w in error.
- Part B: Placebo q2w (Cohort 1[Selected Dose]+Cohort 2): Part B participants exposed to placebo q2w on top of MTX (mean exposure of 40 weeks). 168 participants with inadequate response from Week 16 rescued with high dose of sarilumab (SAR 200 mg q2w) were not included. Excluded 1 participant randomized to placebo q2w who received sarilumab 200 mg q2w in error. He/she was considered in the 200 mg q2w treatment group for safety analysis.
- Part B Sarilumab Rescue: Cohort 1(Selected Doses)+Cohort2: Part B participants exposed to sarilumab 150 mg q2w or 200 mg q2w or placebo q2w, without adequate response from Week 16, rescued with high dose of sarilumab (SAR 200 mg q2w) (mean exposure of 49 weeks from beginning of randomization to the end of rescue treatment).
Arm/Group | Part A: SAR 100 mg qw | Part A: SAR 150 mg qw | Part A: SAR 100 mg q2w | Part A: SAR 150 mg q2w | Part A: SAR 200 mg q2w | Part A: Placebo qw | Part B: SAR 100 mg qw Cohort 1 (Non-selected Dose) | Part B: SAR 150 mg qw Cohort 1 (Non-selected Dose) | Part B: SAR 100 mg q2w Cohort 1 (Non-selected Dose) | Part B: SAR 150 mg q2w (Cohort 1[Selected Dose]+Cohort 2) | Part B: SAR 200 mg q2w (Cohort 1[Selected Dose]+Cohort 2) | Part B: Placebo q2w (Cohort 1[Selected Dose]+Cohort 2) | Part B Sarilumab Rescue: Cohort 1(Selected Doses)+Cohort2
Serious Adverse Events (participants affected / at risk) | 3/50 | 0/50 | 3/51 | 0/52 | 0/51 | 2/51 | 2/29 | 2/26 | 0/29 | 35/370 | 46/369 | 21/259 | 7/284
Other Adverse Events (participants affected / at risk) | 16/50 | 16/50 | 7/51 | 12/52 | 19/51 | 11/51 | 6/29 | 8/26 | 6/29 | 163/370 | 194/369 | 95/259 | 83/284
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: SAR 100 mg qw (N=50) | Part A: SAR 150 mg qw (N=50) | Part A: SAR 100 mg q2w (N=51) | Part A: SAR 150 mg q2w (N=52) | Part A: SAR 200 mg q2w (N=51) | Part A: Placebo qw (N=51) | Part B: SAR 100 mg qw Cohort 1 (Non-selected Dose) (N=29) | Part B: SAR 150 mg qw Cohort 1 (Non-selected Dose) (N=26) | Part B: SAR 100 mg q2w Cohort 1 (Non-selected Dose) (N=29) | Part B: SAR 150 mg q2w (Cohort 1[Selected Dose]+Cohort 2) (N=370) | Part B: SAR 200 mg q2w (Cohort 1[Selected Dose]+Cohort 2) (N=369) | Part B: Placebo q2w (Cohort 1[Selected Dose]+Cohort 2) (N=259) | Part B Sarilumab Rescue: Cohort 1(Selected Doses)+Cohort2 (N=284)
Iron deficiency anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 4 | 0 | 0
Splenic vein thrombosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiovascular insufficiency (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myocardial ischemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Right ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sick sinus syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal wall hematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alcoholic pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Duodenal ulcer hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastric ulcer hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Immediate post-injection reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Impaired healing (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatitis toxic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Abscess oral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Arthritis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0
Bronchitis fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Endometritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Incision site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infected skin ulcer (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Necrotising fasciitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Otitis media acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Otitis media chronic (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pelvic abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0
Pneumonia streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pyelonephritis chronic (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Subacute endocarditis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tinea cruris (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wound hemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Neoplasm of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Embolic cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ischemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Transient ischemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aortic thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Embolism arterial (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Shock hemorrhagic (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: SAR 100 mg qw (N=50) | Part A: SAR 150 mg qw (N=50) | Part A: SAR 100 mg q2w (N=51) | Part A: SAR 150 mg q2w (N=52) | Part A: SAR 200 mg q2w (N=51) | Part A: Placebo qw (N=51) | Part B: SAR 100 mg qw Cohort 1 (Non-selected Dose) (N=29) | Part B: SAR 150 mg qw Cohort 1 (Non-selected Dose) (N=26) | Part B: SAR 100 mg q2w Cohort 1 (Non-selected Dose) (N=29) | Part B: SAR 150 mg q2w (Cohort 1[Selected Dose]+Cohort 2) (N=370) | Part B: SAR 200 mg q2w (Cohort 1[Selected Dose]+Cohort 2) (N=369) | Part B: Placebo q2w (Cohort 1[Selected Dose]+Cohort 2) (N=259) | Part B Sarilumab Rescue: Cohort 1(Selected Doses)+Cohort2 (N=284)
Neutropenia (Blood and lymphatic system disorders) | 6 | 5 | 0 | 1 | 10 | 0 | 1 | 2 | 1 | 36 | 55 | 0 | 5
Injection site erythema (General disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 3 | 0 | 20 | 24 | 2 | 12
Bronchitis (Infections and infestations) | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 12 | 21 | 12 | 7
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 11 | 14 | 3
Nasopharyngitis (Infections and infestations) | 2 | 1 | 2 | 2 | 2 | 3 | 0 | 1 | 0 | 20 | 20 | 12 | 13
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 0 | 2 | 3 | 2 | 0 | 1 | 0 | 31 | 35 | 16 | 14
Urinary tract infection (Infections and infestations) | 3 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 20 | 22 | 10 | 8
Accidental overdose (Injury, poisoning and procedural complications) | 2 | 3 | 1 | 3 | 2 | 5 | 2 | 1 | 3 | 23 | 26 | 17 | 15
Alanine aminotransferase increased (Investigations) | 2 | 2 | 0 | 3 | 2 | 0 | 0 | 1 | 0 | 31 | 30 | 11 | 9
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 10 | 9 | 12
Hypertension (Vascular disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 2 | 2 | 15 | 14 | 10 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.